CLINICAL TRIAL: NCT02102243
Title: The Role of Aldosterone on Sympathetic Nerve Activity and Insulin Sensitivity
Brief Title: Neural Mechanism of Aldosterone-induced Insulin Resistance
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No longer interested in study topic
Sponsor: Wanpen Vongpatanasin (Other)
Responsible Party: Sponsor-Investigator, Wanpen Vongpatanasin, PROFESSOR, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 102010-063
Record Dates: First submitted 2014-03-06; First posted 2014-04-02 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; sympathetic nerve activity; vascular oxidative stress; nitric oxide; nitric oxide synthase (eNOS); endothelium; endothelial dysfunction; endothelial cell protein expression; microvascular blood flow; flow mediated dilation; endothelial cell collection; microbubbles; Definity
MeSH Terms: conditions — Hypertension | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperinsulinemic euglycemic clamp (Experimental): We will perform following procedures:
  DEFINITY® infusion Flow mediated vasodilation Endothelial cell collection Microvascular perfusion assessment using Definity Microneurography
  Interventions: Drug: DEFINITY® infusion; Drug: Human Recombinant Regular Insulin infusion; Drug: Dextrose infusion; Procedure: Flow mediated vasodilation; Procedure: Endothelial cell collection; Procedure: Microvascular perfusion assessment using Definity; Procedure: Microneurography
- Initial Saline Infusion (Experimental): We will perform the following procedures:
  DEFINITY® infusion Human Recombinant Regular Insulin infusion Dextrose infusion Flow mediated vasodilation Endothelial cell collection Microvascular perfusion assessment using Definity Microneurography
  Interventions: Drug: DEFINITY® infusion; Procedure: Flow mediated vasodilation; Procedure: Endothelial cell collection; Procedure: Microvascular perfusion assessment using Definity; Procedure: Microneurography

INTERVENTIONS:
Drug: DEFINITY® infusion — The DEFINITY® vial contains components that upon activation yield perflutren lipid microspheres, a diagnostic drug that is intended to be used for contrast enhancement during echocardiographic procedures. The vial contains a clear, colorless, sterile, non-pyrogenic, hypertonic liquid, which upon activation with agitation, provides a homogeneous, opaque, milky white injectable suspension of perflutren lipid microspheres. The suspension of activated DEFINITY® will be infused intravenously at a rate of 0.20 to 0.27 ml/min, not to exceed a maximum dose of 2 vials per study subject per day or visit.
  Other Names: (IND# 104397)
Drug: Human Recombinant Regular Insulin infusion — The plasma insulin concentration will be acutely raised and maintained at at a steady state by a prime-continuous insulin infusion.
  Other Names: Humulin R; National Drug Code # 0002-8501-01
  Arms: Hyperinsulinemic euglycemic clamp
Drug: Dextrose infusion — The plasma glucose concentration will be held constant at 90 mg/dl by a variable glucose infusion during euglycemic hyperinsulinemic clamp
  Other Names: Dextrose 20%
  Arms: Hyperinsulinemic euglycemic clamp
Procedure: Flow mediated vasodilation — Flow mediated vasodilation (FMD), which is a non-invasive assessment of endothelial function, will be performed on the brachial artery using ultrasound. After a clear picture of the artery has been obtained, the cuff on the same arm will be inflated until it is tight for five minutes. During and following this, the subject's arm will continue to be imaged to monitor maximal increase in the brachial artery diameter.
  Other Names: FMD; Endothelial Dependent Vasodilation
Procedure: Endothelial cell collection — We will collect endothelial cells from a superficial vein, usually in the arm. Following insertion of a peripheral intravenous (IV) catheter, we will collect cells from the inner lining of the vein using a thin, flexible J-tipped wire. The wire will be inserted through the IV into the vein and then removed, along with a sampling of endothelial cells. The cells collected will be processed and stained for several proteins involved in endothelial cell function, using immunofluorescent technique.
Procedure: Microvascular perfusion assessment using Definity — Using high-resolution ultrasound, we will measure skeletal muscle blood flow during infusion of a solution containing the octafluoropropane microbubble contrast agent, Definity. The solution will be a dilution of 1 vial of Definity to 30 cc of normal saline. The ultrasound probe will be placed over the forearm to obtain images while octafluoropropane microbubbles (Definity) are infused intravenously at the rate of 0.20 to 0.27 ml/min, not to exceed a maximum dose of 2 vials per study subject per day or visit. The microvascular perfusion assessment using Definity be performed at rest as well as during slow and fast handgrip exercises.
Procedure: Microneurography — Sympathetic nerve activity from the peroneal nerve measured by inserting a tiny needle directly into the nerve in the leg. Investigators will localize the nerve by electrical stimulation over the skin using a blunt probe. .The recording needle will remain in position throughout the study.
  Other Names: Assessment of sympathetic nerve activity (SNA)

SUMMARY:
Patients with high aldosterone hormone have higher blood glucose than normal people. This study is being done to understand how aldosterone hormone affects the nerve activity that controls blood flow in the muscles and blood glucose. The information may be helpful in selecting blood pressure medications which can improve not only blood pressure but also improve blood sugar.

DETAILED DESCRIPTION:
Patients with primary aldosteronism are known to have impaired insulin sensitivity, which is improved after removal of aldosterone-producing adenoma. In patients with essential hypertension, plasma aldosterone levels have been also shown to positively correlate with indices of insulin resistance.

Mechanism underlying aldosterone-induced insulin resistance is unknown. Aldosterone has been shown to interfere with insulin signaling the vascular cells by increasing production of reactive oxygen species via activation of NADPH oxidase, resulting in decreased availability of nitric oxide (NO), the key mediator for insulin-mediated vasodilation. Treatment with mineralocorticoid receptor antagonists has been shown to improve insulin sensitivity in mice with obesity and metabolic syndrome. Aldosterone has also been shown to increase resting sympathetic vasoconstrictor activity to the peripheral circulation. However, effects of aldosterone and mineralocorticoid receptor antagonists on insulin-mediated skeletal muscle vasodilation, sympathetic activation, and vascular oxidative stress have not been assessed in humans.

The investigators will collect venous endothelial cells, and measure skeletal muscle microvascular perfusion using Octafluoropropane microbubble contrast agents, and measure sympathetic nerve activity in normotensive controls (NT), stage 1 essential hypertensive subjects (ET), and patients with primary aldosteronism (PA) during hyperinsulinemic euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Normotensive controls
2. Stage I (140-159/90-99 mmHg) untreated subjects with essential hypertension
3. Patients with PA and stage I (140-159/90-99 mmHg) hypertension

Exclusion Criteria:

1. Congestive heart failure or coronary artery disease
2. Blood pressure averaging > 159/99 mmHg
3. Serum creatinine > 1.5 mg/dL
4. Diabetes mellitus or other systemic illness
5. Left ventricular hypertrophy by echocardiography or ECG
6. Pregnancy
7. Hypersensitivity to spironolactone, chlorthalidone, amlodipine, human recombinant insulin or Definity
8. Any history of substance abuse (other than tobacco)
9. History of gouty arthritis
10. Patients with right-to-left, bi-directional, or transient right-to-left cardiac shunts
11. Hypersensitivity to perflutren, blood, blood products or albumin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Increase in muscle sympathetic nerve activity during hyperinsulinemic euglycemic clamp | 1 day

SECONDARY OUTCOMES:
Change in microvascular blood flow during hyperinsulinemic euglycemic clamp. | 1 day
Change in microvascular blood flow during saline infusion. | 1 day
Change in endothelial cell protein expression after hyperinsulinemic euglycemic clamp | 1 day
Change in endothelial cell protein expression after saline infusion | 1 day
Increase in muscle sympathetic nerve activity during saline infusion | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Catena C, Lapenna R, Baroselli S, Nadalini E, Colussi G, Novello M, Favret G, Melis A, Cavarape A, Sechi LA. Insulin sensitivity in patients with primary aldosteronism: a follow-up study. J Clin Endocrinol Metab. 2006 Sep;91(9):3457-63. doi: 10.1210/jc.2006-0736. Epub 2006 Jul 5. PMID 16822818
- [Background] Donato AJ, Gano LB, Eskurza I, Silver AE, Gates PE, Jablonski K, Seals DR. Vascular endothelial dysfunction with aging: endothelin-1 and endothelial nitric oxide synthase. Am J Physiol Heart Circ Physiol. 2009 Jul;297(1):H425-32. doi: 10.1152/ajpheart.00689.2008. Epub 2009 May 22. PMID 19465546
- [Background] Colussi G, Catena C, Lapenna R, Nadalini E, Chiuch A, Sechi LA. Insulin resistance and hyperinsulinemia are related to plasma aldosterone levels in hypertensive patients. Diabetes Care. 2007 Sep;30(9):2349-54. doi: 10.2337/dc07-0525. Epub 2007 Jun 15. PMID 17575088
- [Background] Kontak AC, Wang Z, Arbique D, Adams-Huet B, Auchus RJ, Nesbitt SD, Victor RG, Vongpatanasin W. Reversible sympathetic overactivity in hypertensive patients with primary aldosteronism. J Clin Endocrinol Metab. 2010 Oct;95(10):4756-61. doi: 10.1210/jc.2010-0823. Epub 2010 Jul 21. PMID 20660053